CLINICAL TRIAL: NCT02798224
Title: A Post-Visit Patient Portal Tool to Promote Colorectal Cancer Screening
Brief Title: A Patient Portal Tool, E-assist, for Supporting CRC Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: LCCC 1624; 1R01CA197205 (NIH)
Record Dates: First submitted 2016-06-03; First posted 2016-06-14 (Estimated); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer Screening; CRC Screening; Rectum; Colon; Screening; Populations at Risk; CRC; colorectal cancer (CRC)
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- e-assist: Colon Health (treatment arm) (Experimental): Eligible patients identified will receive a prompt (via email) to log into portal for an important health message. Once eligible patient initiates portal session, continuing past IRB consent screen, patient is enrolled.
  Interventions: Behavioral: e-assist: Colon Health
- Healthwise Educational Program (active control) (Active Comparator): Eligible patients identified will receive a prompt (via email) to log into portal for an important health message. Once eligible patient initiates portal session, continuing past IRB consent screen, patient is enrolled.
  Interventions: Behavioral: Healthwise Educational Program
- Usual care control (observational only) (No Intervention): There will be no participant contact in this arm. We will use existing data sources only (e.g., EHRs) to obtain information on participants in this arm (i.e., an observational data review only).

INTERVENTIONS:
Behavioral: e-assist: Colon Health — Online e-assist program uses educational messages and workflow tools. The intent is to reduce mental workload in terms of how to proceed by filtering and presenting information in a usable manner at a time of peaked situational awareness. The program will prompt patients to indicate their decision stage based on the Precaution Adoption Process Model. e-assist users are then prompted to view additional information and logistical assistance personalized for their decision stage.
  Other Names: e-assist; treatment; experimental treatment
  Arms: e-assist: Colon Health (treatment arm)
Behavioral: Healthwise Educational Program — Online access to fact sheets that provide basic information about colorectal cancer and screening.
  Other Names: active control; usual care plus
  Arms: Healthwise Educational Program (active control)

SUMMARY:
To compare patient perceptions, intent to screen, and screening use among those using a patient portal with and without a colorectal cancer (CRC) screening decision support tool, e-assist.

To evaluate whether the effectiveness of e-assist is moderated by multi-level factors, including patient health literacy, decision-making preference, and CRC screening decision stage.

To assess program impact and create an implementation guide for e-assist by combining results from Aims 1 & 2, a program implementation analysis/process evaluation and the perspectives of staff from future diverse implementation sites including small primary care practices, University-based primary practices and federally-qualified health centers.

DETAILED DESCRIPTION:
During initial project period, the content was developed for the online e-assist tool using messages and tools developed under prior NCI-funded applications combined with newly developed messaging specific to this application. Throughout development, the principal investigator will seek input and guidance from a quality improvement team at the Henry Ford Health System (HFHS) (i.e., the local performance site) that is tasked with patient portal innovation for Meaningful Use. Once finalized, the effectiveness of e-assist will be evaluated using a three-arm, practical randomized trial.

Trial participants will be randomized to one of the following three groups:

1. e-assist: Colon Health (treatment arm) [n = 900]
2. Healthwise Educational Program (active control) [n = 900]
3. Usual care control (observational only) [n = 900]

For the evaluation, the investigators employ an intent-to-treat design with primary effectiveness measured by electronic health record (EHR)-documented CRC screening use. Secondary outcomes of interest include patient-reported CRC screening intent, perceived barriers to and support for CRC screening as well as perceived susceptibility and screening benefits. Results from all analyses will be used to develop an implementation guide for the dissemination and implementation of e-assist among diverse primary care practices.

ELIGIBILITY:
Inclusion Criteria:

-CRC screening recommendation via colonoscopy and/or stool cards at time of primary care appointment. Receiving care in a HFHS primary care clinic and activated MyChart account.

Exclusion Criteria:

* EHR-documented colonoscopy in the past 10 years, sigmoidoscopy in the past 5 years, or fecal occult blood test (FOBT) or fecal immunochemical test (FIT) in the past 12 months.
* Elevated risk for CRC (i.e., personal or family history of CRC, those with prior polyps, or a history of inflammatory bowel disease, familial adenomatous polyposis, or hereditary nonpolyposis).

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1826 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2021-07-27 (Actual)

PRIMARY OUTCOMES:
CRC Screening use | 1 year
  For the evaluation, an intent-to-treat design with primary effectiveness measured by electronic health record (EHR)-documented CRC screening use. Effectiveness will be assessed among all trial enrollees and specific subgroups. Primary outcome is a binary variable reflecting CRC screening use at 12-months post-intervention as documented by the occurrence of any of the following: colonoscopy, flexible sigmoidoscopy, fecal occult blood testing, fecal immunochemical testing, or testing via Cologuard.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Elston Lafata, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lafata JE, Shin Y, Flocke SA, Hawley ST, Jones RM, Resnicow K, Schreiber M, Shires DA, Tu SP. Randomised trial to evaluate the effectiveness and impact of offering postvisit decision support and assistance in obtaining physician-recommended colorectal cancer screening: the e-assist: Colon Health study-a protocol study. BMJ Open. 2019 Jan 7;9(1):e023986. doi: 10.1136/bmjopen-2018-023986. PMID 30617102
- [Derived] Dyer KE, Shires DA, Flocke SA, Hawley ST, Jones RM, Resnicow K, Shin Y, Lafata JE. Patient-Reported Needs Following a Referral for Colorectal Cancer Screening. Am J Prev Med. 2019 Feb;56(2):271-280. doi: 10.1016/j.amepre.2018.08.017. Epub 2018 Dec 13. PMID 30554975
- See also: UNC Lineberger Comprehensive Cancer Center — http://unclineberger.org/